CLINICAL TRIAL: NCT07275489
Title: Consequences of Longterm Confinement on Immunity in the Sub-Antarctic Islands : Follow-up of Volunteers on the Kerguelen Islands
Brief Title: CHOICE KERGUELEN 2 : Consequences of Longterm Confinement on Immunity in the Sub-Antarctic Islands : Follow-up of Volunteers on the Kerguelen Islands
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Institut Polaire Français Paul Emile Victor (Unknown)
Responsible Party: Sponsor
Other Study IDs: 49RC25_0439; 2025-A02538-41 (Other: ANSM)
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Human Health in Extreme Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, PBMCs, plasma, serum, urine, saliva, stools, hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HD (healthy donors)
  Interventions: Other: blood ponction; Other: urines collection; Other: hair collection; Other: saliva collection; Other: stools collection

INTERVENTIONS:
Other: blood ponction — blood ponction
Other: urines collection — urines collection
Other: hair collection — hair collection
Other: saliva collection — saliva collection
Other: stools collection — stools collection

SUMMARY:
Living for long periods in extreme environments-like Antarctic research stations or space missions-can have a significant impact on human health, especially on the immune system. Scientists have observed that people in such isolated conditions often experience more infections and a reactivation of viruses that usually stay dormant in the body, such as Herpes viruses. These changes affect both parts of the immune system: the rapid-response "innate" system and the slower, more specific "adaptive" system.

These immune disruptions may be caused by multiple stressors: ongoing psychological stress, disturbed sleep and light cycles (circadian rhythm disruption), and the challenges of living in confined, isolated, and extreme environments. While space missions and Antarctic overwintering programs have provided some insight into these issues, scientists still lack a detailed understanding of how the immune system adapts-or fails to adapt-over time in such conditions.

To help fill this gap, the CHOICE Kerguelen 2 study will follow a group of healthy young adults who will spend one year (from November 2025 to November 2026) in Port-aux-Français, a remote French research station on the Kerguelen Islands in the sub-Antarctic. These volunteers are participating in a civic service program and will be living in a highly isolated environment for the duration of their mission. The CHOICE Kerguelen study is conducted in collaboration with the French Polar Institute (IPEV).

The goal of the study is to collect and store a broad range of biological samples-including blood, saliva, stool, urine, and hair-from these volunteers at four time points during the time of their confinement on the Kerguelent Islands: tevery three months during their stay. These samples will be than analyzed to characterize the immune profiles and intestinal microbiota of the subjects assess eventual viral reactivations and stress biological markers. These analyses will allow to better understand how the immune system reacts to prolonged isolation, and to identify immune profiles that may develop under prolonged stress and limited social contact.

The long-term aim of this project is not only to improve our understanding of human immunity in extreme environments, but also to inform medical research for people living with chronic illness. By studying healthy individuals placed in physically and mentally challenging environments, scientists can better understand how stress and isolation may weaken immune defenses. The findings may one day help design new approaches to support immune health in vulnerable populations.

ELIGIBILITY:
Inclusion Criteria :

* healthy people aged > 18 years
* Participant affiliated with or benefiting from a social security system
* Participant has signed informed consent
* Participant staying as an overwintering member at Kerguelen from November 2025 to November 2026
* Participant included in the CELREMED research project of the University Hospital of Angers on helathy volunteers in the context of CHOICE Kerguelen 1 protocol

Exclusion Criteria:

* age < 18 years
* Pregnant, breastfeeding, or postpartum woman
* immunocompromised people (primary immunodeficiency, HIV infection or immunosupressive treatment)
* Person refusing to participate in the study
* Person with a history of autoimmune disease - -Person deprived of liberty by judicial or administrative decision
* Person undergoing involuntary psychiatric treatment
* Person subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participant included in the CELREMED research project of the University Hospital of Angers on helathy volunteers in the context of CHOICE Kerguelen 1 protocol
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
lymphocytes subsets during overwintering on the Kerguelen Islands | At inclusion (3 months after the beginning of overwintering)
  lymphocytes subsets by flow cytometry
lymphocytes subsets during overwintering on the Kerguelen Islands | At 3 months (6 months after the beginning of overwintering )
  lymphocytes subsets by flow cytometry
lymphocytes subsets during overwintering on the Kerguelen Islands | At 6 months (9 months after the beginning of overwintering )
  lymphocytes subsets by flow cytometry
lymphocytes subsets during overwintering on the Kerguelen Islands | At 9 months (12 months after the beginning of overwintering )
  lymphocytes subsets by flow cytometry
RNAsep during overwintering on the Kerguelen Islands | At inclusion (3 months after the beginning of overwintering )
  RNAseq
RNAsep during overwintering on the Kerguelen Islands | At 3 months (6 months after the beginning of overwintering )
  RNAseq
RNAsep during overwintering on the Kerguelen Islands | At 6 months (9 months after the beginning of overwintering )
  RNAseq
RNAsep during overwintering on the Kerguelen Islands | At 9 months (12 months after the beginning of overwintering )
  RNAseq
plasmatic cytokines during overwintering on the Kerguelen Islands | At inclusion (3 months after the beginning of overwintering )
  plasmatic cytokines by Bioplex
plasmatic cytokines during overwintering on the Kerguelen Islands | At 3 months (6 months after the beginning of overwintering )
  plasmatic cytokines by Bioplex
plasmatic cytokines during overwintering on the Kerguelen Islands | At 6 months (9 months after the beginning of overwintering )
  plasmatic cytokines by Bioplex
plasmatic cytokines during overwintering on the Kerguelen Islands | At 9 months (12 months after the beginning of overwintering )
  plasmatic cytokines by Bioplex
fecal microbiota | At inclusion (3 months after the beginning of overwintering )
  fecal microbiota by bacterial sequencing
fecal microbiota | At 3 months (6 months after the beginning of overwintering )
  fecal microbiota by bacterial sequencing
fecal microbiota | At 6 months (9 months after the beginning of overwintering )
  fecal microbiota by bacterial sequencing
fecal microbiota | At 9 months (12 months after the beginning of overwintering )
  fecal microbiota by bacterial sequencing
hormonal stress markers during overwintering on the Kerguelen Islands | At inclusion (3 months after the beginning of overwintering )
  hormonal stress markers assessment in blood/urinary/hair by Elisa and nephelemetry
hormonal stress markers during overwintering on the Kerguelen Islands | At 3 months (6 months after the beginning of overwintering )
  hormonal stress markers assessment in blood/urinary/hair by Elisa and nephelemetry
hormonal stress markers during overwintering on the Kerguelen Islands | At 6 months (9 months after the beginning of overwintering )
  hormonal stress markers assessment in blood/urinary/hair by Elisa and nephelemetry
hormonal stress markers during overwintering on the Kerguelen Islands | At 9 months (12 months after the beginning of overwintering )
  hormonal stress markers assessment in blood/urinary/hair by Elisa and nephelemetry
stress profile during overwintering on the Kerguelen Islands | At inclusion (3 months after the beginning of overwintering )
  psychological stress by CST test form
stress profile during overwintering on the Kerguelen Islands | At 3 months (6 months after the beginning of overwintering )
  psychological stress by CST test form
stress profile during overwintering on the Kerguelen Islands | At 6 months (9 months after the beginning of overwintering )
  psychological stress by CST test form
stress profile during overwintering on the Kerguelen Islands | At 9 months (12 months after the beginning of overwintering )
  psychological stress by CST test form

SECONDARY OUTCOMES:
EBV viral reactivations during overwintering on the Kerguelen Islands | At inclusion (3 months after the beginning of overwintering )
  EBV in blood and saliva by quantitative PCR
EBV viral reactivations during overwintering on the Kerguelen Islands | At 3 months (6 months after the beginning of overwintering )
  EBV in blood and saliva by quantitative PCR
EBV viral reactivations during overwintering on the Kerguelen Islands | At 6 months (9 months after the beginning of overwintering )
  EBV in blood and saliva by quantitative PCR
EBV viral reactivations during overwintering on the Kerguelen Islands | At 9 months (12 months after the beginning of overwintering )
  EBV in blood and saliva by quantitative PCR
CMV viral reactivations during overwintering on the Kerguelen Islands | At inclusion (3 months after the beginning of overwintering )
  CMV in blood and saliva by quantitative PCR
CMV viral reactivations during overwintering on the Kerguelen Islands | At 3 months (6 months after the beginning of overwintering )
  CMV in blood and saliva by quantitative PCR
CMV viral reactivations during overwintering on the Kerguelen Islands | At 6 months (9 months after the beginning of overwintering )
  CMV in blood and saliva by quantitative PCR
CMV viral reactivations during overwintering on the Kerguelen Islands | At 9 months (12 months after the beginning of overwintering )
  CMV in blood and saliva by quantitative PCR
HSV viral reactivations during overwintering on the Kerguelen Islands | At inclusion (3 months after the beginning of overwintering )
  HSV in blood and saliva by quantitative PCR
HSV viral reactivations during overwintering on the Kerguelen Islands | At 3 months (6 months after the beginning of overwintering )
  HSV in blood and saliva by quantitative PCR
HSV viral reactivations during overwintering on the Kerguelen Islands | At 6 months (9 months after the beginning of overwintering )
  HSV in blood and saliva by quantitative PCR
HSV viral reactivations during overwintering on the Kerguelen Islands | At 9 months (12 months after the beginning of overwintering )
  HSV in blood and saliva by quantitative PCR
TTV viral reactivations during overwintering on the Kerguelen Islands | At inclusion (3 months after the beginning of overwintering )
  TTV viral loads in blood and saliva by quantitative PCR
TTV viral reactivations during overwintering on the Kerguelen Islands | At 3 months (6 months after the beginning of overwintering )
  TTV viral loads in blood and saliva by quantitative PCR
TTV viral reactivations during overwintering on the Kerguelen Islands | At 6 months (9 months after the beginning of overwintering )
  TTV viral loads in blood and saliva by quantitative PCR
TTV viral reactivations during overwintering on the Kerguelen Islands | At 9 months (12 months after the beginning of overwintering )
  TTV viral loads in blood and saliva by quantitative PCR

CONTACTS AND LOCATIONS:
Overall Officials: Charline MIOT, MD, Principal Investigator — University Hospital, Angers
Locations (1):
- Hôpital SAMUKER, Port-aux-français/ Archipel KERGUELEN /Terres Australes et Antarctiques Françaises, Port-aux-Français, Terres Australes Et Antarctiques Françaises, French Southern and Antarctic Lands

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).